CLINICAL TRIAL: NCT04784858
Title: Integrating a Parenting Intervention Into Substance Use Treatment: A Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Niagara Health System (Other); house of sophrosyne (Unknown)
Responsible Party: Principal Investigator, Karen Milligan, Associate Professor, Toronto Metropolitan University
Other Study IDs: ABCforECD
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Parenting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While motherhood is central to the design of maternal integrated substance use treatment programs, "evidence-based" parenting interventions tailored to the needs of the population are rare. Stakeholder engagement has revealed that the evidence-base is not reflective of the needs of client population. With 34 ECD programs in Ontario, ECD programs are unique position to pilot Attachment and Biobehavioral Catch Up (ABC) and see if it is a good fit for their clients and if it is effective and feasible. ABC is 10-week evidence-based parenting intervention for parents who live in the context of complex risk, including mental health, addictions, child welfare involvement, and poverty. Investigators of this project will complete a open label mixed method feasibility pilot study involving active implementation of ABC that will involve: 1. exploration facilitators and barriers of the year-long implementation and training process and 2. exploration of changes in maternal mental health, substance use and parenting outcomes from beginning to end of treatment. Results of this mixed method pilot study will inform a larger trial with a control group and support a funding application to support its completion.

DETAILED DESCRIPTION:
While motherhood is central to the design of maternal integrated substance use treatment programs, there are few "evidence-based" parenting interventions tailored to the needs of the population. This study will address this limitation in current parenting intervention research by exploring if Attachment and Biobehavioral Catch Up (ABC) is well suited and feasible to implement within integrated maternal substance use outpatient treatment. ABC is 10-week evidence-based parenting intervention for parents who live in the context of complex risk, including mental health, addictions, child welfare involvement, and poverty. Investigators of this project will complete a open label mixed method feasibility pilot study involving active implementation of ABC that will involve: 1. exploration facilitators and barriers of the year-long implementation and training process and 2. exploration of changes in maternal mental health, substance use and parenting outcomes from beginning to end of treatment. Results of this mixed method pilot study will inform a larger trial with a control group and support a funding application to support its completion.

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant/parenting children ages 6-24 months
* Women that are clients of participating ECD agencies

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers who experience vulnerability and are challenged by substance use disorder trauma, and/or poverty.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Maternal Sensitivity | 9 minutes play session
  Coded from observed parent-child interactions

SECONDARY OUTCOMES:
Reflective Functioning | 5 minutes
  Reflective Function (RF) 18-item questionnaire
Parental Reflective Functioning | 5 minutes
  Reflective Function Questionnaire (PRF-Q) 8-item questionnaire
Depression, Anxiety, and Stress | 8 minutes
  Depression, Anxiety and Stress Scale (DASS21) - 21 item questionnaire
Parenting Stress | 10 minutes
  Parental Stress Index (PSI) - Short Form, 36 item questionnaire
Perceived Social Support | 5 minutes
  Multidimensional Scale of Perceived Social Support (MSPS), 12 item questionnaire
Difficulties in Emotion Regulation | 5 minutes
  Difficulties in Emotion Regulation Scale-SF (DERS-SF), 18-item questionnaire
Substance use screener | 2 minutes
  Global Appraisal of Individual Needs (Substance Use) (GAIN), 5-item questionnaire
Interpersonal Emotion Regulation | 8 minutes
  Interpersonal Emotion Regulation Questionnaire (IERQ), 20-item

CONTACTS AND LOCATIONS:
Overall Officials: Karen Milligan, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No